CLINICAL TRIAL: NCT04288375
Title: Reduction of Dose and Volume in Postoperative Radiation for Extremity Soft Tissue Sarcoma
Brief Title: Dose Reduction of Postoperative Radiation for Soft Tissue Sarcoma of the Arms and Legs
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-064
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Soft Tissue Sarcoma
Keywords: Postoperative Radiation; Soft Tissue Sarcoma of extremity; 20-064
MeSH Terms: conditions — Sarcoma | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- extremity soft tissue sarcoma (STS) (Experimental): Postoperative radiation therapy to the primary site with a reduction in radiation dose and volume. Specifically, the tumor bed plus a margin of 2cm craniocaudally and 1.5cm radially will be utilized to create the clinical target volume. The total dose will consist of 50 Gy in 25 fractions.
  Interventions: Radiation: Intensity-modulated radiation therapy (IMRT)

INTERVENTIONS:
Radiation: Intensity-modulated radiation therapy (IMRT) — The prescribed dose of radiations for all patients will be 50 Gy in 25 fractions. 6MV energy photons will be used. Multi-beam IMRT plans, utilizing dynamic multileaf collimation, will be created based on the target tissue coverage and normal tissue avoidance.

SUMMARY:
The investigators are doing this study to find out whether lowering the dose of postoperative radiation therapy and targeting a smaller area of tissue for treatment is as effective as the standard dose and volume of radiation therapy to control soft tissue sarcoma after surgery. They also want to find out whether the study approach causes fewer and less severe long-term side effects than the standard approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with a primary soft tissue sarcoma of the extremity, confirmed by MSKCC pathologic review
* Age at the time of enrollment of ≥18 years
* Patients must have undergone margin-negative oncologic resection of their primary tumor, as confirmed by MSKCC pathologic review
* Patients must be able to start radiation within 3 months from time of surgery

  °If patient is receiving adjuvant chemotherapy, patient must start RT no longer than 3 months past their chemo treatment.
* Female patients of childbearing potential must have a negative serum pregnancy test within 14 days of radiation start (or if urine test, within 24 hours of radiation start)
* Sexually active patients of childbearing potential must agree to use effective contraception.
* The use of chemotherapy will not be dictated by this trial. Patients are allowed to receive chemotherapy at the discretion of the disease management team (as is standard practice to make individualized decisions for each patient regarding the use of chemotherapy).

Exclusion Criteria:

* Patients with positive margins after surgical resection as indicated by MSKCC pathologic review
* Patients with diagnosis of superficial myxofibrosarcoma with indistinct/infiltrative borders on preoperative MRI16 (see Appendix Figure 1 for reference figure)
* Patients with multifocal disease in the extremity
* Patients who have received prior radiotherapy at or adjacent to the primary tumor bed
* Patients with a differentinvasive cancer requiring active treatment at the time of enrollment.
* Patients with any concurrent medical or psychiatric condition or disease which, in the investigator's judgment, would make them inappropriate candidates for entry into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-26 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of local control at 2 years. | 2 years
  will be assessed via imaging of the primary tumor site (MRI preferred, CT for patients who cannot get or tolerate an MRI). Imaging must take place at least annually for the first two years post-radiation. Local failure is defined as a relapse in the primary tumor bed.

SECONDARY OUTCOMES:
overall survival | 2 years
  will be performed for each patient using clinical data obtained from chart review 2 years after the last patient enrolled is treated. Will use Kaplan Meier methods to estimate survival at 2 years after RT starting at the end of RT

CONTACTS AND LOCATIONS:
Overall Officials: Kaled Alektiar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All protocol activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (All protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All protocol activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm